CLINICAL TRIAL: NCT03124550
Title: Development of An Exergame for Caregivers of Individuals With Alzheimer's Disease or Related Dementias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Margie Lachman, Professor of Psychology, Brandeis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Exergame #17065; 5P30AG048785 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Sedentary Lifestyle; Stress, Psychological
Keywords: Caregivers; Exercise; Behavior Change
MeSH Terms: conditions — Sedentary Behavior; Stress, Psychological; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will use the exergame for 6 weeks. Physical activity will be recorded. Participants will receive game-related rewards when they are active.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exergame Experience (Experimental): Participants will use the exergame for 6 weeks, during which time game telemetry data (all interactions with the software) will be automatically logged by the system. The participants will be asked to use the game at least every other day. Caregivers will be sent an email or text message to remind them to use the system if they have not done so within three days. Utilizing two-way text messaging, an experience sampling protocol will be employed: once per week, participants will be sent brief questions probing their level of satisfaction with the exergame and their level of perceived connectedness to the community of other caregivers using the exergame.
  Interventions: Behavioral: Exergame Experience

INTERVENTIONS:
Behavioral: Exergame Experience — Fitbit Charge HR will be used to measure physical activity and sedentary behavior during waking hours. Each participant will wear a Fitbit for a period of one week at baseline and during the entire 6-week pilot study. Data on step counts, heart rate, and moderate/vigorous activity from the Fitbits will be transmitted wirelessly to our secure research server and will be used to assess changes in physical activity and sedentary behavior over the course of the study. Participants will be instructed to wear the monitor continuously on the wrist. Data will be analyzed using previously validated accelerometer count cut-points for adults after accounting for invalid data and wear time.

SUMMARY:
The study goal is to evaluate user experience with our developed exergame, which was designed to increase physical activity, exercise self-efficacy, and social connections among caregivers of individuals with Alzheimer's disease (AD) or related dementias. Participants will use this garden-themed exergame for six weeks. Tailoring an exergame for caregivers of AD or related dementias has the potential to increase physical activity and to improve overall health and well-being in this vulnerable population, which in turn can benefit the patients for whom they provide care. All study sessions be held at a location convenient to participants.

DETAILED DESCRIPTION:
The number of Alzheimer's Disease (AD) caregivers providing informal care for family members is rising dramatically, and supportive programs are vitally needed. Caregivers of AD patients have relatively high levels of stress and depression and limited physical activity and social engagement. Technology-driven programs can offer engaging, sustainable, and scalable opportunities to give caregivers critically-needed supports for health and well- being. This pilot study uses cognitive behavioral methods to develop an innovative social exergame to increase physical and social activity among AD caregivers. Leveraging wearable activity monitors, physical activity data collected throughout the day and in varied settings will serve as input to the game experience.

Caregivers will assess the suitability of an exergame prototype with an array of features including (1) instructional exercise modules, (2) activity data visualizations, (3) digital rewards for physical activity that can be used to create virtual gardens, and (4) opportunities to connect virtually with other caregivers to share and comment on their creative products.

The aim of this study is to evaluate enjoyment of the exergame and its feasibility to increase moderate and vigorous physical activity, virtual social contact, and exercise self-efficacy. A group of approximately 20 caregivers will test the exergame for six weeks on an Android smartphone. The findings will be used to develop larger-scale intervention studies to test the efficacy of the exergame in the future. Tailoring an exergame for caregivers of AD has the potential to increase physical activity and to improve overall health and well-being in this vulnerable population, which in turn can benefit the Alzheimer's patients for whom they provide care.

All participants will be given a fitness tracker to keep after the study, a value of over $100! Participants will receive $5 Amazon Gift card each week upon completion of each weekly questionnaire. Participants can receive up to a $30 of Amazon Gift card upon completion of weekly questionnaire.

ELIGIBILITY:
Inclusion criteria:

* Be 18 years or older
* Be a caregiver who spends a significant amount of time with a family member, partner, or friend with Alzheimer's Disease or related dementias.
* Be able to walk for at least 20 minutes at a time
* Have regular access to an Android smartphone with Internet access
* Be comfortable wearing a fitness tracker for the duration of the study
* Must be located in Massachusetts, New Hampshire, Rhode Island, Connecticut, or New York City

Exclusion Criteria:

* A recent (within the past 6 months) cardiovascular event or fall.
* A score on the Short Portable Mental Status Questionnaire (SPMSQ) that indicates intellectual impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margie Lachman, Ph.D., Principal Investigator — Brandeis University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exergame Experience
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exergame Experience
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18
Education [Count of Participants; unit: Participants]
  Less Than 7th Grade | 0
  Junior high/middle school | 0
  Some high school | 2
  Completed high school or GED | 4
  Some college or Vocational training | 1
  Completed 2 years of college, Associate Degree | 1
  Completed 4 years college, College Degree | 7
  Completed graduate school degree | 3
Care Recipient [Count of Participants; unit: Participants]
  Parent | 10
  Other family members | 6
  Friend | 2
Age of Care Recipient [Mean (Standard Deviation); unit: years] | 80 (8)
Caregiving Length [Mean (Standard Deviation); unit: Months] | 45 (33)
Caregiving Time [Mean (Standard Deviation); unit: Days per Week] | 5 (2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Steps
Description: Number of steps recorded daily from the Fitbit, weekly step averages
Time Frame: Daily for six weeks
Population: Daily step averages less than 500 steps were classified as a missing day of data. Weekly step averages were calculated for weeks with 4 or more days of valid data.
Measure: Mean (Standard Deviation); unit: Daily Steps
Arm/Group | Exergame Experience
Number analyzed (Participants) | 18
Daily Steps
  Week 1 | 8857 (5132)
  Week 2 | 8179 (4263)
  Week 3 | 8659 (5280)
  Week 4 | 7867 (5428)
  Week 5 | 6554 (4301)
  Week 6 | 6837 (4413)
Statistical Analysis 1: Comparison: Exergame Experience; Multilevel modeling with the LMER package in R was used to determine whether participants changed in weekly average steps over the 6-week intervention; Test type: Other; p = .0008, Multilevel Modeling

2. Secondary Outcome: Caregiver's Management of Distress
Description: Caregiver's management of distress was measured with the amount of time caregivers spent on themselves doing leisure activities when they were under stress from caregiving. Answer choices ranged from never (1) to very often (4). A higher score indicated better management of distress.
Time Frame: Baseline (pretest) and 6 weeks from the start of the intervention (posttest)
Population: Because of participant family emergencies, one of the participant did not get to complete the posttest. Therefore, we missed the pre and post test comparison for one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exergame Experience
Number analyzed (Participants) | 17
units on a scale
  Pre-test | 2.1 (.39)
  Post-test | 2.4 (.30)
Statistical Analysis 1: Comparison: Exergame Experience; Pre-test and post-test comparison; Test type: Superiority; p = .01, t-test, 2 sided

3. Secondary Outcome: Exercise Self-efficacy
Description: A modified version of Bandura's Exercise Self-Efficacy scale (Bandura, 1997) was used in the current study. This 8-item scale assesses how sure one is that they would exercise under different conditions or constraints (e.g. How sure are you that you will exercise when you are feeling down or depressed?), with answer choices ranging from not sure at all (1) to very sure (4). The 8 items are averaged to create a composite score, where a higher score indicates greater exercise self-efficacy (Neupert et al., 2009).
Time Frame: Baseline (pretest) and 6 weeks from the start of the intervention (posttest)
Population: Because of participant family emergencies, one of the participant did not get to complete the posttest. Therefore, we missed the pre and post test comparison for one participant. Another participant did not fill out the pretest for the exercise self-efficacy section. Thus, we only analyzed 16 participants for exercise self-efficacy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exergame Experience
Number analyzed (Participants) | 16
units on a scale
  Pre-test | 2.59 (1.02)
  Post-test | 2.61 (1.06)
Statistical Analysis 1: Comparison: Exergame Experience; Pre-test and post-test comparison; Test type: Superiority; p = .94, t-test, 2 sided

4. Secondary Outcome: Number of Social Contacts
Description: Average daily number of social contacts with other caregivers using the exergame in a week
Time Frame: Daily for six weeks
Population: Social contact is measured daily by the sum of number of times participants viewed, liked, added, and replied to stories, and viewed other caregivers' gardens.
Measure: Mean (Standard Deviation); unit: Daily number of social contact
Arm/Group | Exergame Experience
Number analyzed (Participants) | 18
Daily number of social contact
  Week 1 | 5.7 (7.4)
  Week 2 | 4.8 (5.0)
  Week 3 | 4.7 (5.1)
  Week 4 | 3.7 (4.6)
  Week 5 | 3.9 (7.2)
  Week 6 | 3.4 (6.2)
Statistical Analysis 1: Comparison: Exergame Experience; Multilevel modeling with the LMER package in R was used to determine whether participants changed in weekly number of social contact over the 6-week intervention; Test type: Other; p = .0007, Multilevel Modeling

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Participants were asked to report any adverse events to the investigator throughout the study
Arm/Group | Exergame Experience
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-03-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03124550/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03124550/Prot_SAP_001.pdf